CLINICAL TRIAL: NCT02572258
Title: The Effect of Supplementary Food Cookies on Prevention of Moderate Malnutrition in Preschool Children in Rural Mexico
Brief Title: Supplementary Food on Prevention of Moderate Malnutrition in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-1410
Record Dates: First submitted 2015-09-29; First posted 2015-10-08 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Moderate Acute Malnutrition (MAM)

ARMS (2):
- Nutritional oats cookie and educational session (Experimental): Nutritional cookie with oats and nuts
  Interventions: Other: Nutritional cookie
- Educational session only (No Intervention)

INTERVENTIONS:
Other: Nutritional cookie
  Arms: Nutritional oats cookie and educational session

SUMMARY:
The study will evaluate the impact of a supplementary food (cookies) in preventing the risk of developing moderate acute malnutrition (MAM) in preschool mildly malnourished children.

Children will be divided in two groups; one will received the cookie plus 12 educative sessions and the other just the educative program. The study will last 12 months

ELIGIBILITY:
Inclusion Criteria:

* (2-5 years old), who are from low socioeconomic classes (E and D classes)
* reside in rural areas, and with WHZ- between > -3 and ≤ -2, and
* informed consent given by the subject's mother or caregiver

Exclusion Criteria:

* Severe acute malnutrition (HAZ, WAZ and WHZ-scores ≤-3) based on the 2006 World Health Organization (WHO) reference values (24)
* Vitamin A deficiency (softening, ulceration, cloudiness of the cornea, and dryness of the conjunctivitis), and iodine deficiency (visible goiter)
* (3 or more episodes of loose/liquid stools/per day and lasted more than 24-hours), fever (high temperature that lasted more than 24 hours as reported by the mother/caregiver), and respiratory infections (coughing and/or runny nose that last more than 24 hours).
* Current consumption of other supplementary foods.
* Peanut or other ingredient allergy based on prior report. If some direct family member is allergic to peanuts, child would not be enrolled.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1048 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Weight (kg) for height (cm) Z-score | 12 months

SECONDARY OUTCOMES:
Weight (kg) gains | 12 months
height (cm) for age (months) Z-score | 12 months
weight (kg) for age (months) Z-score | 12 months
Mid-upper arm circumference (cm) (MUAC) | 12 months
height (cm) gains | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Juan Talavera, PhD, Principal Investigator — Universidad Autónoma del Estado de México
Locations (1):
- Un Kilo de Ayuda, Colonia Lomas de Chapultepec, Mexico City, Mexico